CLINICAL TRIAL: NCT06084182
Title: The Relationship Between Cognitive Function and Functional Capacity, Cognitive Reserve, Reaction Time in Patients With Multiple Sclerosis
Brief Title: Cognitive Function in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/2611
Record Dates: First submitted 2022-11-18; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; cognitive function; cognitive reserve; functional capacity
MeSH Terms: conditions — Multiple Sclerosis | interventions — Reaction Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Other): Patients with a definite diagnosis of MS according to McDonald diagnostic criteria
  Interventions: Other: Cognitive function, cognitive reserve, functional capacity, reaction time, strength, fatigue, depression and general health assessment
- Control Group (No Intervention): Healthy individuals

INTERVENTIONS:
Other: Cognitive function, cognitive reserve, functional capacity, reaction time, strength, fatigue, depression and general health assessment — 6-minute walk test and 5-time sit-to-stand test (STS-5) were used for functional capacity assessment. For cognitive reserve assessment, the Cognitive Reserve Index questionnaire was used. Reaction time, cognitive function and visiospatial perception were evaluated with the mobile application. In addition, the Fatigue Severity Scale; Beck Depression Questionnaire and Nottingham Health Profile were used.
  Arms: Patient group

SUMMARY:
The aim of the study is to investigate the relationship between cognitive function, functional capacity, cognitive reserve and reaction time in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Cognitive impairment in patients with MS is a common problem that significantly affects quality of life. It shows an association between functional capacity and physical fitness levels and cognition in non-MS populations, and especially in the elderly.

Although cognitive dysfunctions are known, few studies have been found on its relationship with secondary problems caused by the disease and its correlation with other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS diagnosis
* Expanded Disability Status Scale score <5.5
* Being able to use a smart phone
* No relapse during the last 30 days
* Being between the ages of 18-65
* Mini-Mental State Examination score>24

Exclusion Criteria:

* Severe Visual Impairment
* Severe Psychiatric Disorder,
* Severe Arthritis in Knee or Hip,
* Pregnancy and other neurological or vestibular disorders that may prevent the patient from completing the functional examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Functional capacity assessment | Baseline
  6-minute walk test were used. The 6-minute walk test requires patients to cover as much distance as possible in a six-minute period. The walking distance is recorded.
Functional capacity assessment | baseline
  The STS-5 test, on the other hand, requires patients to perform five sit-stand cycles in a standard chair (0.43-m high and 0.45-m wide) as quickly as possible, measured in seconds, and is used as an indicator of lower extremity muscle strength.
Cognitive function | Baseline
  A mobile application called Trail Making Test was used to evaluate visual attention and cognitive flexibility. The completion time of subsections A and B was recorded. Working memory will be evaluated using a mobile application called Digit Span test. This application gives your maximum digit memory. This score has been saved.
Visiospatial perception | Baseline
  The visuospatial perception was evaluated with the help of the mobile application called Corsi Block Tapping test. The highest span in this application is recorded.
Cognitive Reserve Index Questionnaire | Baseline
  A tool used to quantify, in a standardized model, cognitive reserve through an interview to the participant or to the caregiver. The questionnaire collects demographic information regarding the school curriculum, work and type of free-time activities. These three different indices (CRI-School, CRI-Work and CRI-Free Time) are then combined into a single "Index of Cognitive Reserve".

SECONDARY OUTCOMES:
Hand grip strength | Baseline
  Handgrip was measured with the Baseline Digital Hand Dynamometer 135 KG®. The results were recorded as Kg.
Nottingham Health Profile. | Baseline
  Nottingham Health Profile consists of 6 sections and a total of 38 questions evaluating patients' pain, emotional reaction, sleep, social isolation, physical activity and energy. In this questionnaire, where the highest score is 600 points, a high score is associated with a deterioration in quality of life
Beck Depression Inventory | Baseline
  The Beck Depression Inventory is a self-report measure of depression severity that is a well-characterized scale with excellent psychometric properties and is frequently used in research studies of depression.
  The scale measures symptoms related to sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping pattern, irritability, changes in appetite, concentration difficulty, tiredness or fatigue, and loss of interest in sex.
  We report the total score on the Beck Depression Inventory, which has a range of 0 to 63. Higher values represent greater severity of depression. The following score interpretations are provided in the scale's manual:
  0-9 minimal depression 10-18 mild depression 19-29 moderate depression 30-63 severe depression
Fatigue Severity Scale. | Baseline
  The fatigue severity scale is a short measurement tool consisting of nine questions developed by Krupp and used to measure the degree of fatigue in patients with multiple sclerosis. The validity and reliability of the scale Armutlu et al. and Cronbach's alpha coefficient was found to be 0.94. In the scale, individuals are asked to rate the fatigue they have felt during the past week from 1 to 7. Each section is scored between 1 (strongly disagree) and 7 (strongly agree). The total score is calculated by taking the average of nine items.
Reaction time | Baseline
  A mobile application called "Tap fast" was used. The patient is asked to touch the maximum number of boxes by touching the screen as quickly as possible within 15 seconds. The patient's score was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Engin Ramazanoglu, Study Chair — Inonu University; Mehmet Tecellioglu, Study Chair — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

REFERENCES:
- [Derived] Candiri B, Ramazanoglu E, Talu B, Tecellioglu M. The relationship between cognitive function and functional capacity, and cognitive reserve and reaction time in patients with multiple sclerosis. Arq Neuropsiquiatr. 2024 Sep;82(9):1-9. doi: 10.1055/s-0044-1788273. Epub 2024 Aug 26. PMID 39187267